CLINICAL TRIAL: NCT00738400
Title: Double-blind, Placebo Controlled, Randomized Study of Vardenafil to Determine Efficacy on Erectile Dysfunction (ED) in Men With ED and Metabolic Syndrome (ED-METABOLIC)
Brief Title: Study of Vardenafil in Patients Suffering From Erectile Dysfunction and Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13171; 2008-002140-41 (EudraCT Number); ED-METABOLIC (Other: Company Internal)
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Results first posted 2011-06-01 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Erectile Dysfunction; Metabolic Syndrome
Keywords: Vardenafil; Erectile Dysfunction; Double-blind study
MeSH Terms: conditions — Erectile Dysfunction; Metabolic Syndrome | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vardenafil (Levitra, BAY38-9456) (Experimental): Vardenafil 10 mg tablets PRN (pro re nata) for 4 weeks, Vardenafil 5 mg/10 mg/20 mg tablets PRN for consecutive 4 weeks
  Interventions: Drug: Vardenafil (Levitra, BAY38-9456)
- Placebo (Placebo Comparator): Matching placebo tablets PRN (pro re nata) for 4 weeks, placebo tablets PRN for consecutive 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil (Levitra, BAY38-9456) — Vardenafil 10 mg tablets daily for 4 weeks, vardenafil 5 mg / 10 mg / 20 mg tablets for consecutive 4 weeks
  Arms: Vardenafil (Levitra, BAY38-9456)
Drug: Placebo — Matching placebo tablets daily for 4 weeks, placebo tablets daily for consecutive 4 weeks
  Arms: Placebo

SUMMARY:
This is a controlled, randomized, multi-center prospective study of vardenafil to determine efficacy on Erectile Dysfunction (ED), tolerability and safety in men with ED and Metabolic Syndrome. This study will explore the rate of patients who do need to switch to the highest dosage based upon the expectation that most men can stay on vardenafil 10 mg PRN (pro re nata)

ELIGIBILITY:
Inclusion Criteria:

* Stable heterosexual relationship
* History of erectile dysfunction for at least 6 months
* IIEF- EF Domain entry score (at Visit 2): >21 points
* Documented metabolic syndrome according to the IDF (International Diabetes Foundation)
* Subjects motivated for erectile dysfunction treatment
* Documented, dated, written informed consent

Exclusion Criteria:

* Any underlying cardiovascular condition
* History of myocardial infarction
* Uncontrolled atrial fibrillation
* Resting hypotension
* Postural hypotension within 6 months of Visit 1
* History of congenital QT prolongation
* Bleeding disorder
* History of prostatectomy because of prostate cancer
* Hereditary degenerative retinal disorders
* History of loss of vision because of NAION (non-arteritic anterior ischemic optic neuropathy)
* 29 Additional Exclusion Criteria

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (18):
- Germany (18):
  - Cham, Bavaria
  - Regensburg, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Stuhr, Lower Saxony
  - Bonn, North Rhine-Westphalia
  - Grevenbroich, North Rhine-Westphalia
  - Leverkusen, North Rhine-Westphalia
  - Mülheim, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Dierdorf, Rhineland-Palatinate
  - Koblenz, Rhineland-Palatinate
  - Trier, Rhineland-Palatinate
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
  - Berlin, State of Berlin

REFERENCES:
- [Result] Schneider T, Gleissner J, Merfort F, Hermanns M, Beneke M, Ulbrich E. Efficacy and safety of vardenafil for the treatment of erectile dysfunction in men with metabolic syndrome: results of a randomized, placebo-controlled trial. J Sex Med. 2011 Oct;8(10):2904-11. doi: 10.1111/j.1743-6109.2011.02383.x. Epub 2011 Jul 19. PMID 21771281
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Started | 76 | 74
Received Treatment, Safety Population | 75 (One invalid participant (no evidence that this randomized participant took study medication).) | 72 (Two invalid participants (no evidence that these randomized participants took study medication).)
ITT (Intent To Treatment) Population | 75 | 70 (No post-baseline efficacy measurement in 2 participants)
Completed | 72 | 67
Not Completed | 4 | 7
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Non-compliant with study medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo | Total
Number analyzed (Participants) | 75 | 72 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] — Number of participants analyzed for baseline (visit 2) was safety population.
  years | 56.3 (5.9) | 55.6 (6.7) | 56.0 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants analyzed for baseline (visit 2) was safety population.
  Participants
    Female | 0 | 0 | 0
    Male | 75 | 72 | 147
BMI (body mass index) [Mean (Standard Deviation); unit: kg/m^2] — Number of participants analyzed for baseline (visit 2) was safety population.
  kg/m^2 | 30.4 (3.6) | 30.4 (3.4) | 30.4 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Index of Erectile Function - Erectile Function Domain (IIEF-EF) Subscore at Week 8 or Last Observation Carried Forward (LOCF)
Description: The primary variable was the least square (LS)-mean difference between treatment groups in the IIEF-EF domain score (6-30 ordinal points, specifying the severity of erectile dysfunction: 6-10 'severe'; 11-16 'moderate'; 17-21 'mild to moderate'; 22-25 'mild'; 26-30 'no erectile dysfunction [ED]'). The target variable is the LS-mean difference between treatment groups at endpoint. The LS-means of both treatment groups are derived from a baseline-adjusted endpoint measure (week 8/last observation carried forward [LOCF]) as calculated via an ANCOVA.
Time Frame: baseline and up to 8 weeks or LOCF
Population: Number of participants analyzed differs due to missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 74 | 70
Scores on a scale | 20.96 [19.38 to 22.54] | 14.20 [12.57 to 15.83]
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; ANCOVA, baseline covariate, endpoint week 8 or LOCF. Factors: treatment, pooled centers. Ls mean at endpoint; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -6.76, 95% CI [-9.03 to -4.49]

2. Primary Outcome: Change in Percentage From Baseline in Success of Penetration (SEP2: Sexual Encounter Profile Question 2) at Week 8
Description: Percent successful penetrations were calculated per participant as the number of successful sexual attempts (penetrations) divided by the total number of attempts. The mean percent successful penetrations was then calculated across all participants.
Time Frame: Baseline and 8 weeks
Population: Number of participants analyzed differs due to missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent successful penetrations
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 73 | 64
Percent successful penetrations | 73.50 [66.71 to 80.30] | 52.79 [45.51 to 60.08]
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; ANCOVA, baseline covariate, endpoint week 8 or LOCF. Factors: treatment, pooled centers. Ls mean at endpoint; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -20.71, 95% CI [-30.66 to -10.76]

3. Primary Outcome: Change in Percentage From Baseline in Success of Erection Maintenance (SEP3: Sexual Encounter Profile Question 3) at Week 8
Description: Percent successful maintenance of erection were calculated per participant as the number of successful attempts (maintenance of erection) divided by the total number of attempts. The mean percent successful maintenance of erection was then calculated across all participants.
Time Frame: Baseline and 8 weeks
Population: Number of participants analyzed differs due to missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent erection maintenance
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 73 | 64
Percent erection maintenance | 53.15 [45.42 to 60.89] | 27.00 [18.70 to 35.29]
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; ANCOVA, baseline covariate, endpoint week 8 or LOCF. Factors: treatment, pooled centers. Ls mean at endpoint; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -26.16, 95% CI [-37.48 to -14.83]

4. Secondary Outcome: Percentage of Participants Achieving "Back to Normal" Erectile Function at Week 8 or Last Observation Carried Forward (LOCF)
Description: Responders: percentage of participants achieving an IIEF-EF score >25.(IIEF-EF domain score: 6-30 ordinal points, specifying the severity of erectile dysfunction: 6-10 'severe'; 11-16 'moderate'; 17-21 'mild to moderate'; 22-25 'mild'; 26-30 'no ED')
Time Frame: up to 8 weeks or LOCF
Population: Number of participants analyzed differs due to missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 74 | 70
Percentage of participants | 35 | 10
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; Mantel-Haenszel Test; Test type: Superiority or Other; p = 0.0004, Mantel Haenszel

5. Secondary Outcome: Change in Percentage From Baseline in Ability to Obtain an Erection (SEP1) at Week 8
Description: Percent successful erections were calculated per participant as the number of successful attempts (achievement of erection) divided by the total number of attempts. The mean percent successful erections was then calculated across all participants.
Time Frame: Baseline and 8 weeks
Population: Number of participants analyzed differs due to missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent successful erections
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 73 | 64
Percent successful erections | 91.36 [85.74 to 96.97] | 75.79 [69.76 to 81.81]
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; ANCOVA, baseline covariate, endpoint week 8 or LOCF. Factors: treatment, pooled centers. Ls mean at endpoint; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -15.57, 95% CI [-23.80 to -7.34]

6. Secondary Outcome: Change in Percentage From Baseline in Ability to Ejaculate (SEP6) at Week 8
Description: Percent successful ejaculations were calculated per participant as the number of successful attempts (achievement of ejaculation) divided by the total number of attempts. The mean percent successful ejaculations was then calculated across all participants.
Time Frame: Baseline and 8 weeks
Population: Number of participants analyzed differs due to missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent successful ejaculations
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 73 | 64
Percent successful ejaculations | 71.29 [64.53 to 78.06] | 43.96 [36.71 to 51.21]
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; ANCOVA, baseline covariate, endpoint week 8 or LOCF. Factors: treatment, pooled centers. Ls mean at endpoint; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -27.33, 95% CI [-37.24 to -17.43]

7. Secondary Outcome: Number of Participants Who Can Stay on the Initially Provided Dosage of Vardenafil (10 mg PRN (Pro re Nata))
Description: Number of participants with no recorded titration of Vardenafil after visit 3.
Time Frame: week 4 and week 8
Measure: Number; unit: Participants
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 75 | 70
Participants | 28 | 13

ADVERSE EVENTS:
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/72
Other Adverse Events (participants affected / at risk) | 16/75 | 8/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vardenafil (Levitra, BAY38-9456) (N=75) | Placebo (N=72)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Balanitis candida (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (13) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Premature ejaculation (Psychiatric disorders) | 1 (1) | 0 (0)
Balanitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (4) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less